CLINICAL TRIAL: NCT02198898
Title: Prospective Multicenter Trial for Anti-adhesion Effect of GUARDIX-SGⓇ Following Radical Gastrectomy in Patients With Gastric Cancer.
Brief Title: Anti-adhesion Effect of GUARDIX-SGⓇ in Gastric Cancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kyo Young Song, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUMCGC1301; GUARDIXGASTRIC (Other: The Catholic University of Korea)
Record Dates: First submitted 2013-06-29; First posted 2014-07-24 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Adhesive Intestinal Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GUARDIX (No Intervention): no guadix
- guadix (Experimental): guadix treatment
  Interventions: Device: GUARDIX-SG

INTERVENTIONS:
Device: GUARDIX-SG
  Arms: guadix

SUMMARY:
This study is to evaluate the efficacy of GUARDIX-SGⓇ for patients with gastrectomy in Korea and the investigators hypothesized applying of adhesive preventing agent would reduce incidence of adhesive obstruction after gastrectomy.

DETAILED DESCRIPTION:
Adhesive bowel obstruction is relatively often complication in patients after abdominal surgery

Gastric cancer is the most frequent cancer in Korea.

The incidence of adhesive bowel obstruction would be increased in patients with gastric cancer, especially associated radical lymphadenectomy.

The causes of postoperative adhesive obstruction include adhesion of the wound, adhesion of small intestine to small intestine, adhesion of the small intestine to other abdominal organs, and internal hernia.

Several studies reported efficacy of adhesive preventing agent after colorectal resection.

Gastrectomy is associated with a high risk (incidence, 11.7%-38.5%) of bowel obstruction.

To date, however, no randomized study has shown that GUARDIX-SGⓇ reduces the rate of small bowel obstruction after gastrectomy with radical lymphadenectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric adenocarcinoma who scheduled to undergo open gastrectomy
* Informed consents

Exclusion Criteria:

* Pregnant
* Ascites
* Liver dysfunction
* Renal failure
* Past history of abdominal operation or small bowel obstruction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
incidence of adhesive intestinal obstruction | up to 1 years after operation (every 3 month)
  the incidence of adhesive bowel obstruction between using GUARDIX-SG group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Young Song, M.D., Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea